CLINICAL TRIAL: NCT05494840
Title: The Effect of Prenatal Haptonomy on Pregnancy-related Anxiety, Distress and Psychological Well-being
Brief Title: The Effect of Prenatal Haptonomy on Anxiety, Distress and Psychological Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Özbek (Other)
Responsible Party: Sponsor-Investigator, Hilal Özbek, Assist. Prof. Dr, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TR TOKAT01
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: First Pregnancy
Keywords: haptonomy; distress; psychological well-being; anxiety
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Haptonomy- first experimental Group (Experimental): Haptonomy Group Pregnant school will made to the experimental group, and haptonomy will be applied for at least 30 minutes, once a week for 6 weeks (with the researcher).
  Interventions: Behavioral: Haptonomy
- Haptonomy- second experimental Group (Experimental): Haptonomy Group Pregnant school will made to the experimental group, and haptonomy will be applied for at least 30 minutes, once a week for 3 weeks (with the researcher).
  Interventions: Behavioral: Haptonomy
- Haptonomy- Control Group (No Intervention): Standard of care Group The control group will not be interfered with.

INTERVENTIONS:
Behavioral: Haptonomy — Haptonomy, as a field dealing with emotional contact through touch, describe the relationship between parents and the unborn baby.
  Arms: Haptonomy- first experimental Group; Haptonomy- second experimental Group

SUMMARY:
Introduction:Anksiyete experienced during prenatal can increase Distress, cause negative perinatal outcomes, and adversely affect the psychological well-being. This study will conducted to determine the effect of prenatal haptonomy on pregnancy-related anxiety, distress and psychological well-being.

Methods: The population of the randomized controlled experimental study will consist of 102 primiparous pregnant women within the gestational weeks 22-27 who presented to the pregnant school of a state hospital in Turkey (34 first experimental group, 34 second experimental group, 34 control group).

DETAILED DESCRIPTION:
Background: Anksiyete experienced during prenatal can increase Distress, cause negative perinatal outcomes, and adversely affect the psychological well-being.

Aim: This study will conducted to determine the effect of prenatal haptonomy on pregnancy-related anxiety, distress and psychological well-being.

Metod: For the educational study of the research, the midwife working in the Pregnant Class will be interviewed and informed about it. The mat and seat cushions in the Pregnant Class will be arranged by the researcher in a way that is suitable for the application. Music will be played during the application. Wellness music recommended by the haptonomy trainer will be selected for the music (Rathfisch, 2019). Haptonomy application is planned to be performed individually with pregnant women. Pregnant women in the experimental group 1 and 2 will be given the haptonomy application together with the trainings (standard care practices) in the pregnant class, and the pregnant women in the control group will only be trained in the pregnant class. Pregnant class trainings include reproductive health physiology, problems that can be seen in pregnancy, birth process, newborn care, covering the prenatal period, birth and postpartum period.

Haptonomy- first experimental Group: Haptonomy Group Pregnant school will made to the experimental group, and haptonomy will be applied for at least 30 minutes, once a week for 6 weeks (with the researcher).

Haptonomy- second experimental Group: Haptonomy Group Pregnant school will made to the experimental group, and haptonomy will be applied for at least 30 minutes, once a week for 3 weeks (with the researcher).

Haptonomy- Control Group: Standard of care Group The control group will not be interfered with.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women who were married,
* aged 18 years and over,
* literate,
* living in the city center,
* not having any health problems in themselves and their infants,
* with spontaneous pregnancy at 22-27 weeks of gestation,
* without perception and communication problems,
* and who agreed to participate in the study were included in the study.

Exclusion Criteria:

• Multiparity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy-Related Anxiety Questionnaire-Revised-2 (PRAQ-R2) | Baseline
  This scale consisting of 10 items is a 5-point Likert-type scale to question women's pregnancy-related anxiety levels. The scale items are scored between 1 and 5 (1-Absolutely not relevant and 5-Very relevant). The lowest and highest scores are 11 and 55 for primiparous women, and 10 and 50 for multiparous women, respectively. A higher scale score indicates a higher level of anxiety in pregnancy.
Tilburg Pregnancy Distress Scale (TPDS) | Baseline
  This scale consisting of 16 items is a 4-point Likert-type scale. The scale items are scored between 0 and 3 (very often 0 points, quite often 1 point, occasionally 2 points, rarely/never 3 points). A total score of 28 and above according to the cut-off point indicates that the pregnant woman is at risk for distress.
Psychological well-being scale | Baseline
  This scale consisting of 8 items is a 7-point Likert-type scale. The scale items are scored between 1 and 7 (1-Absolutely not relevant and 7-Very relevant). The lowest and highest scores are 8 and 56 respectively. A high score indicates that the person has many psychological resources and strengths.

SECONDARY OUTCOMES:
Pregnancy-Related Anxiety Questionnaire-Revised-2 (PRAQ-R2) | Week 3
  This scale consisting of 10 items is a 5-point Likert-type scale to question women's pregnancy-related anxiety levels. The scale items are scored between 1 and 5 (1-Absolutely not relevant and 5-Very relevant). The lowest and highest scores are 11 and 55 for primiparous women, and 10 and 50 for multiparous women, respectively. A higher scale score indicates a higher level of anxiety in pregnancy.
Tilburg Pregnancy Distress Scale (TPDS) | Week 3
  This scale consisting of 16 items is a 4-point Likert-type scale. The scale items are scored between 0 and 3 (very often 0 points, quite often 1 point, occasionally 2 points, rarely/never 3 points). A total score of 28 and above according to the cut-off point indicates that the pregnant woman is at risk for distress.
Psychological well-being scale | Week 3
  This scale consisting of 8 items is a 7-point Likert-type scale. The scale items are scored between 1 and 7 (1-Absolutely not relevant and 7-Very relevant). The lowest and highest scores are 8 and 56 respectively. A high score indicates that the person has many psychological resources and strengths.

OTHER OUTCOMES:
Pregnancy-Related Anxiety Questionnaire-Revised-2 (PRAQ-R2) | Week 6
  This scale consisting of 10 items is a 5-point Likert-type scale to question women's pregnancy-related anxiety levels. The scale items are scored between 1 and 5 (1-Absolutely not relevant and 5-Very relevant). The lowest and highest scores are 11 and 55 for primiparous women, and 10 and 50 for multiparous women, respectively. A higher scale score indicates a higher level of anxiety in pregnancy.
Tilburg Pregnancy Distress Scale (TPDS) | Week 6
  This scale consisting of 16 items is a 4-point Likert-type scale. The scale items are scored between 0 and 3 (very often 0 points, quite often 1 point, occasionally 2 points, rarely/never 3 points). A total score of 28 and above according to the cut-off point indicates that the pregnant woman is at risk for distress.
Psychological well-being scale | Week 6
  This scale consisting of 8 items is a 7-point Likert-type scale. The scale items are scored between 1 and 7 (1-Absolutely not relevant and 7-Very relevant). The lowest and highest scores are 8 and 56 respectively. A high score indicates that the person has many psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Özbek, Principal Investigator — Tokat Gaziosmanpaşa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Adam, E. M. (2012). L ' haptonomie Un projetpourunenaissance [Un projetpourunenaissance]. Université Henri Poincaré, Nancy I.
- [Background] Aksoy Derya Y, Timur Tashan S, Duman M, Durgun Ozan Y. Turkish adaptation of the pregnancy-related anxiety questionnaire-revised 2: Validity and reliability study in multiparous and primiparous pregnancy. Midwifery. 2018 Jul;62:61-68. doi: 10.1016/j.midw.2018.03.006. Epub 2018 Mar 27. PMID 29655006
- [Background] Arabin, B., & Metz, G. A. S. (2020). Environmental enrichment and pregnancy: Paradigms of (epi)genetic effects of social or sensory stimulation. Gynakologe, 53(7), 433-443. https://doi.org/10.1007/s00129-020-04622-2
- [Background] Bilgen, O., & Tekim, U. (2020). Marriage Satisfaction In Thelast Three Months Of Pregnancy The Effect On Depression. USBED, 2(2), 138153.
- [Background] Capik A, Pasinlioglu T. Validity and reliability study of the Tilburg Pregnancy Distress Scale into Turkish. J Psychiatr Ment Health Nurs. 2015 May;22(4):260-9. doi: 10.1111/jpm.12211. PMID 25912270
- [Background] Célestin-Lhopiteau, I., & Wanquet-Thibault, P. (2018). Haptonomie. In Guide des pratiques psychocorporelles: 25 techniques (relaxation, hypnoseart-thérapie, toucher, etc.) (2nd ed., pp. 186-190). Elsevier Health Sciences.
- [Background] Çiltaş, N. Y., & Köse Tuncer, S. (2019). Gebelikte Distresin Tanımlanması: Erzincan Örneği. Mehmet Akif Ersoy Üniversitesi Sağlık Bilimleri Enstitüsü Dergisi, 7(1), 15-24. https://doi.org/10.24998/maeusabed.518546
- [Background] CIRDH. (2018). Haptonomie pré et postnatale. International Center for Research and Development of Haptonomy. https://www.haptonomie.org/fr/espace-public/accompagnement-haptonomique-pre-et-postnatal.html
- [Background] Dufay, L. (2019). École de Psychologues Praticiens [Mémoire De Recherche en vue de l'obtention du Diplôme De Psychologue, École de Psychologues Pratıcıens Instıtut Catholıque de Parıs].
- [Background] Duman M, Durgun Ozan Y, Aksoy Derya Y, Timur Tashan S. The effect of relaxation exercises training on pregnancy-related anxiety after perinatal loss: A pilot randomized control trial✰. Explore (NY). 2022 Jan-Feb;18(1):44-50. doi: 10.1016/j.explore.2020.11.002. Epub 2020 Nov 17. PMID 33229283
- [Background] Hulsbosch LP, Nyklicek I, Potharst ES, Meems M, Boekhorst MGBM, Pop VJM. Online mindfulness-based intervention for women with pregnancy distress: design of a randomized controlled trial. BMC Pregnancy Childbirth. 2020 Mar 13;20(1):159. doi: 10.1186/s12884-020-2843-0. PMID 32169030
- [Background] Kaya Zaman, F., Ozkan, N., & Toprak, D. (2018). Depression and Anxiety in Pregnancy. Konuralp Medical Journal, 10(1), 20-25. https://doi.org/10.18521/ktd.311793
- [Background] Kilic, A., & Can Gürkan, Ö. (2021). Evidence-Based Use of Music Therapy During Pregnancy, Birth and Postpartum. KTO Karatay University Journal of Health Sciences. 2(1): 47-60.
- [Background] Klabbers, G. A. (2018). Can haptotherapy reduce fear of childbirth? Some first answers from a randomized controlled trial [PhD Thesis]. Tilburg Üniversity.
- [Background] Paica, C. I. (2017). Prenatal and Postnatal Psychological Counselling The conscious assumption of the maternal role. Journal of Experiential Psychotherapy, 20(2), 24-31.
- [Background] Rathfisch, Gulay. (2019). Prenatal haptonomy course notes [PowerPoint slide]. İstanbul.
- [Background] Simsek Kucukkelepce, D., Aydin Ozkan, S., & Yilmaz, S. (2022). Investigation of the relationship between postpartum depression in primiparous pregnants experiencing psychological distress during pregnancy: Prospective study. Journal of Social and Analytical Health, 2(1), 8-14. https://doi.org/10.5281/ZENODO.6342685
- [Background] Telef, B. B. (2011). The Adaptation of Psychological Well-Being into Turkish: A Validity and Reliability Study. XI. Psychological Counseling and Guidance Congress.
- [Background] Telef, B. B. (2013). The Adaptation of Psychological Well-Being into Turkish: A Validity and Reliability Study. HU Journal of Education, 28(3), 374-384.
- [Background] Veldman F. Philosophy behind science. Confirming affectivity, the dawn of human life: the pre-, peri- and postnatal affective-confirming. Haptonomic accompaniment of parents and their child. Neuro Endocrinol Lett. 2001 Aug;22(4):295-304. PMID 11524636
- [Background] Yan H, Ding Y, Guo W. Mental Health of Pregnant and Postpartum Women During the Coronavirus Disease 2019 Pandemic: A Systematic Review and Meta-Analysis. Front Psychol. 2020 Nov 25;11:617001. doi: 10.3389/fpsyg.2020.617001. eCollection 2020. PMID 33324308